CLINICAL TRIAL: NCT02986893
Title: Pilot Study of a Dietary Intervention for Multiple Sclerosis (MS)
Brief Title: Pilot Diet Study for Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 16-0288
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Diet; Clinical Trial
MeSH Terms: conditions — Multiple Sclerosis | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Intervention Arm (Experimental): Participants will be assigned to follow a specific dietary intervention for 6 months
  Interventions: Behavioral: Dietary Intervention
- Non-dietary Intervention Arm (Experimental): Participants will continue their usual diet and will be invited to attend monthly meetings at the MS Center for 6 months
  Interventions: Behavioral: Non-dietary Intervention Arm

INTERVENTIONS:
Behavioral: Dietary Intervention — Participants will be assigned to follow a specific diet for 6 months. This will involve meetings with the study nutritionist at least monthly as well as regular assessments related to adherence and effects.
  Arms: Dietary Intervention Arm
Behavioral: Non-dietary Intervention Arm — Participants will be requested to follow their usual diet and attend monthly meetings at the MS center to discuss various topics with a focus on wellness in MS for 6 months.
  Other Names: Monthly MS Center meeting attendance
  Arms: Non-dietary Intervention Arm

SUMMARY:
The goal of this project is to establish the feasibility of dietary research in Multiple Sclerosis (MS) patients as well as to provide preliminary data to support future clinical trials of diet in MS. This project is a pilot randomized trial of a dietary intervention in MS patients. The dietary intervention was designed to include dietary components that have been suggested to be of benefit in MS through basic science research and observational-type studies in MS patients and to exclude those that have been suggested to be detrimental. It is therefore rich in foods that are high in polyunsaturated fatty acids (particularly omega-3 fatty acids), foods that are high in polyphenols and antioxidant vitamins such as berries and other fruits and vegetables, as well as whole grains, and excludes meat other than fish as well as dairy and refined sugars and limits salt. Subjects are randomly assigned to the dietary intervention or to the non-intervention group. The non-intervention group will be invited to attend regular meetings with a focus on wellness in MS however will not receive specific dietary instructions. At the end of the study those who were not in the dietary intervention group will have the opportunity to receive all of the materials used during the study should they wish to begin the diet.

DETAILED DESCRIPTION:
This is a pilot study of a carefully-designed dietary intervention that aims to help overcome obstacles to diet research in MS as well as provide needed preliminary data for future clinical trials. It incorporates elements with suggested benefits for MS including foods high in polyunsaturated fatty acids, polyphenols, and antioxidants, and excludes those that are potentially detrimental such as dairy and saturated fat from meat, refined sugars, and also limits salt content.

The 15 participants randomized to the dietary intervention arm will undergo intensive training with a nutritionist and the PI regarding the mechanics of the diet. Menu suggestions, recipes, and grocery lists will be provided. This will be followed by regular meetings and contact with all study participants by e-mail and phone to maximize dietary adherence. The 15 subjects not in the dietary intervention group will have regular meetings at the center with a focus on wellness in MS in general. Adherence to the diet will be assessed through the use of multiple validated dietary questionnaires as well as through biological specimen analysis. Feedback will be requested to provide valuable advice from participants that can be applied to future clinical trials. Effects on general health and wellness outcomes such as BMI, lipid profile, fasting glucose, hemoglobin a1c, blood pressure, as well as effects on fatigue and cognition will be explored. Fecal specimens for microbiota analysis and blood samples for immunological profiling will be collected and stored for future analysis to help elucidate potential mechanisms for dietary effects.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65, inclusive
* Female
* Self-reported race of white or black
* Diagnosis of CIS with MRI consistent with MS, RRMS, or PPMS by McDonald 2010 criteria or SPMS by Lublin 2014 definition
* If the subject is receiving treatment with disease-modifying therapy, must be on that therapy for at least 3 months prior to randomization
* Willing and able to be randomized to dietary intervention with commitment to rigorously follow the dietary protocol and complete the necessary assessments over 6 months

Exclusion Criteria:

* MS exacerbation within 60 days of protocol start
* Intravenous corticosteroids within 60 days of protocol start
* Patients with severe medical or psychiatric illness that would interfere with their ability to comply with the protocol, or potentially cause the patient harm as determined by the treating physician
* Active smoking at the time of protocol start
* Taking supplements other than approved doses of vitamin D within 1 month of study start
* Pregnancy or planning pregnancy during the study period, breastfeeding

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-11; Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Food Frequency Questionnaire | at 6 months
  Adherence to the dietary intervention will be assessed through the food frequency questionnaire. This full-length (approximately 110 food item) questionnaire was designed to estimate usual and customary intake of a wide array of nutrients and food groups. Calculations are estimated via computerized software programs.
Carotenoids level | at 6 months
  Adherence to the dietary intervention assessed through the carotenoid biological marker.
Pooled fatty acids level | at 6 months
  Adherence to the dietary intervention assessed through the pooled fatty acids biological marker.
Urinary sodium level | at 6 months
  Adherence to the dietary intervention assessed through the urinary sodium biological marker.

SECONDARY OUTCOMES:
Change in Blood pressure | Baseline, 3 months, 6 months
  Change in Blood pressure at 3 months and 6 months as compared to baseline
Change in body mass index | Baseline, 3 months, 6 months
  Change in body mass index at 3 months and 6 months as compared to baseline
Change in lipid profile | Baseline, 6 months
  Change in lipid profile at 6 months as compared to baseline
Change in fasting glucose level | Baseline, 6 months
  Change in fasting glucose at 6 months as compared to baseline
Change in hemoglobin a1c level | Baseline, 6 months
  Change in hemoglobin a1c at 6 months as compared to baseline
Change in Multiple Sclerosis Impact Scale-29 (MSIS-29) | Baseline, 3 months, 6 months
  Change in quality of life questionnaire scores as assessed by the Multiple Sclerosis Impact Scale-29 at 3 months and 6 months as compared to baseline. The MSIS-29 is a new measure of the physical and psychological impact of MS from the patient's perspective. Each item is scored from 1 (not at all) to 5 (extremely), with total scale from 29 to 145.
Change in Multiple Sclerosis Quality of Life-54 (MSQOL-54) | Baseline, 3 months, 6 months
  Change in quality of life questionnaire scores as assessed by the Multiple Sclerosis Quality of Life-54 questionnaire at 3 months and 6 months as compared to baseline. The MSQOL-54 is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. There is no single overall score for the MSQOL-54. The MSQOL-54 items are transformed linearly to 0-100 scores and final scores are obtained by averaging items within the scales. Two summary scores - physical health and mental health - can be derived from a weighted combination of scale scores.
Change in the Minimum Assessment of Cognitive Function in MS (MACFIMS) | Baseline, 6 months
  Change at 6 months from baseline. Total range of MACFIMS from 0 (severe impairment to 282 (severe impairment) which is composed of 7 neuropsychological tests: 1) Controlled Oral Word Association Test (COWAT) score 0 (nonverbal) to 22 (normal verbal fluency; 2) Judgment of Line Orientation (JLO) score 0 (no visuospatial skills) to 30 (normal visuospatial skills); 3) California Verbal Learning Test, 2nd ed (CLVT-II) score 0 (severe deficit) to 16 (normal recall); 4) Brief Visuospatial Memory Test-Revised (BVMT-R) score 0 (poor visuospatial memory) to 12 (normal visuospatial memory); 5) Paced Auditory Serial Addition Test (PASAT) score 0 (poor cognitive function) to 60 (normal cognitive function); 6) Delis-Kaplan Executive Function System (DKEFS) score 0 (poor cognitive function) to 32 (higher levels of creative and abstract thought ); and 7) Symbol Digit Modalities Test (SDMT) score 0 (neurological impairment) to 110 (no impairment ).
Neurological Fatigue Index-MS | Baseline, 6 months
  Change in fatigue scale score (Neurological Fatigue Index-MS) at 6 months as compared to baseline. The Neurological Fatigue Index is a 9 item questionnaire with each item scored 1 (not appropriate) to 7 (agree). The score is calculated by the average response to the questions (adding up all the answers and dividing by 9). full range from 1 to 9 with higher value indicating more fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Katz Sand, MD, Principal Investigator — Corinne Goldsmith Dickinson Center for Multiple Sclerosis at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No